CLINICAL TRIAL: NCT00800839
Title: Busulfan (IV) and Fludarabine Followed by Post-allogeneic Transplantation Cyclophosphamide for Graft-versus-Host Disease Prophylaxis in Patients With Hematologic Malignancies.
Brief Title: Busulfan and Fludarabine Followed by Post-transplant Cyclophosphamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0261; NCI-2012-01660 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Hematologic Diseases; Leukemia; Lymphoma; Myeloma
Keywords: Post-allogeneic transplantation; Graft-versus-Host Disease Prophylaxis; Graft-versus-Host Disease; GVHD; Hematologic malignancies; Leukemia; Lymphoma; Myeloma; Human Leukocyte Antigen; HLA; Busulfan; Cyclophosphamide; Fludarabine; Mesna; Cytoxan®; Neosar®; Busulfex; Myleran®; Fludarabine Phosphate
MeSH Terms: conditions — Hematologic Diseases; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Graft vs Host Disease; Hematologic Neoplasms | interventions — Busulfan; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Busulfan + Fludarabine + Cyclophosphamide (Experimental): Busulfan starting dose of 32 mg/m^2 by vein over 3 hours each day. Test dose day -8 (inpatient) or test dose day -30 to day -8 (outpatient) and then, days -6,-5,-4, and -3. Fludarabine dose of 40 mg/m^2 by vein over 1 hour each day on Day -6 through Day -3 before receiving Busulfan. Cyclophosphamide dose of 50 mg/kg by vein over 3 hours on Days 3 and 4.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Busulfan — Starting dose of 32 mg/m^2 by vein over 3 hours each day. Test dose day -8 (inpatient) or test dose day -30 to day -8 (outpatient) and then, days -6,-5,-4, and -3.
  Other Names: Bulsulfex™; Myleran®
Drug: Fludarabine — Dose of 40 mg/m^2 by vein over 1 hour each day on Day -6 through Day -3 before receiving Busulfan.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Cyclophosphamide — Dose of 50 mg/kg by vein over 3 hours on Days 3 and 4.
  Other Names: Cytoxan®; Neosar®

SUMMARY:
The goal of this clinical research study is to learn if cyclophosphamide given after busulfan and fludarabine can help to prevent graft versus host disease (GVHD - a condition in which transplanted tissue attacks the body into which it is transplanted) in patients receiving a stem cell transplant. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Busulfan is designed to bind to DNA (the genetic material of cells), which may cause cancer cells to die.

Fludarabine is designed to make cancer cells less able to repair damaged DNA. This may increase the likelihood of the cells dying.

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die. It is also designed to suppress the immune system and help prevent GVHD.

Study Drug Administration and Transplant:

If you are an inpatient, on Day -8 (8 days before the date of transplant), you will receive a low-level test dose of busulfan through a needle in your vein over 1 hour.

If you are an outpatient, on Day -30 through Day -8, you will receive a low-level test dose of busulfan through a needle in your vein over 1 hour each day.

You will be given an anti-seizure drug to help prevent seizures each time you receive busulfan. Your doctor will explain how the drug will be given and the drug's risks. Seizures are a rare but serious side effect of busulfan.

On Days -8, -6, and -4, blood (about 1 teaspoon each time) will then be drawn a total of 11 times for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points. This PK testing will be done to find the dose of busulfan needed for your body size on the other days that you receive busulfan.

On Day -6 through Day -3, you will receive your body-specific dose of busulfan by vein over 3 hours each day. If you cannot have the blood level tests performed for any reason, you will receive the standard busulfan dose. You will receive fludarabine through a needle in your vein over 1 hour on each of these days before you receive busulfan.

On Day 0, you will receive the donor bone marrow or blood stem cells by vein over about 1 hour.

On Day +3 and Day +4, you will receive cyclophosphamide by vein over 3 hours.

On Days +3 thru +5 just before the first dose of cyclophosphamide and then every 4 hours, you will receive mesna by vein over 30 minutes for a total of 10 doses. Mesna is a drug that protects bladder cells from damage by chemotherapy drugs. It is used to decrease the risk of bleeding in the bladder.

Once a day starting on Day +7, you will receive filgrastim (G-CSF -- a drug that helps with the growth of white blood cells) through a needle under your skin until your blood cell levels reach "recovered" levels for 3 days in a row.

Study Visits:

Every day you are in the hospital and at each outpatient visit, you will have a physical exam to check for symptoms of GVHD.

Blood (about 3 teaspoons) will be drawn at least 2 times a week for the first 100 days after the transplant for routine tests.

About 1 month after your transplant, then once every 3 months up to a year, the following tests and procedures will be performed:

* Blood (about 5 tablespoons) will be drawn for routine tests and to check for CMV. Blood draws may be repeated more often, if you doctor thinks it is needed.
* Urine will be collected for routine tests.
* You will have a bone marrow aspirate and biopsy to check the status of the disease.

At Months 1, 2, 3, 6, and 12 after your transplant, blood (about 4 tablespoons) will be drawn to check the status of your immune system.

Tests and procedures may be repeated more often during the study, if your doctor thinks it is needed.

Length of Study:

You will be on study in the hospital for about 4 weeks. You will be taken off study if the disease gets worse or if the study doctor thinks it is in your best interest.

Long-Term Follow-Up:

After the first 24 months, you will receive either a phone call or a letter from the study doctor or your regular doctor 1 time each year to check the status of the disease. If you are contacted by mail, you will be given a self-addressed stamped envelope with which you can return your responses to the doctor.

This is an investigational study. Busulfan is FDA approved and commercially available for the treatment of chronic myelogenous leukemia (CML). Fludarabine is FDA approved and commercially available for the treatment of chronic lymphocytic leukemia (CLL). Cyclophosphamide is FDA approved and commercially available for the treatment of lymphoma. The use of these drugs together for the possible prevention of GVHD is investigational.

Up to 40 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high risk hematological malignancies, including those with induction failure and after treated or untreated relapse.
2. HLA-identical sibling or matched unrelated donor transplants not eligible for protocols of higher priority.
3. Age 6 months to 75 years.
4. Bilirubin </= 1.5 mg/dl, serum glutamate pyruvate transaminase (SGPT) </= 200 IU/ml (unless Gilbert's syndrome).
5. Calculated creatinine clearance of >50mL/min using the Cockcroft-Gault equation for adult patients 18 to 70 years old, and the Schwartz equation for pediatric patients 6 months to 17 years old.
6. Diffusing capacity for carbon monoxide (DLCO) >45% predicted corrected for hemoglobin (as reported by the Pulmonary Function Laboratory at MDACC). For most children </= 6 years of age who are unable to perform pulmonary function test (PFT), pulse oximetry >/= 92% on room air.
7. left ventricular ejection fraction (LVEF) >/= 35%.

Exclusion Criteria:

1. HIV seropositivity
2. Uncontrolled infections.
3. Positive Beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization
4. Inability to sign consent

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-09; Primary Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amin Alousi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 02, 2008 to December 12, 2011. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Started | 56
Completed | 49
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 61 [39 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Grade II to IV Acute GVHD
Description: Graft Versus Host Disease (GVHD) defined as grade 2 to 4 GVHD within first 100 days post transplant. Death or disease progression before diagnosis of GVHD were considered competing risks in the estimation of the incidence of acute GVHD.
Time Frame: 100 days post transplant
Measure: Number (95% Confidence Interval); unit: percentage of incidence
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 49
percentage of incidence | 53 [40 to 70]

2. Primary Outcome: Cumulative Incidence of Grade III to IV Acute GVHD
Description: Graft Versus Host Disease (GVHD) defined as grade 3 to 4 GVHD within first 100 days post transplant. Death or disease progression before diagnosis of GVHD were considered competing risks in the estimation of the incidence of acute GVHD.
Time Frame: 100 days post transplant
Measure: Number (95% Confidence Interval); unit: percentage of incidence
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 49
percentage of incidence | 22 [13 to 38]

3. Primary Outcome: Day-100 Treatment-Related Mortality
Description: Treatment-Related Mortality (TRM) was estimated from the date of transplant using the cumulative incidence method to account for competing risks. Disease progression or relapse death were considered competing risk for TRM.
Time Frame: 100 days post transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 49
percentage of participants | 14 [7 to 28]

4. Secondary Outcome: Rate of Engraftment
Description: Engraftment defined as the evidence of donor derived cells (more than 5%) by bone marrow chimerism studies in the presence of neutrophil recovery by day 28 post stem cell (SC) infusion. Engraftment date is the first day of three (3) consecutive days that the ANC exceeds 0.5 x109/L. Delayed engraftment is defined as the evidence of engraftment beyond day 28 post SC infusion achieved after the administration of therapeutic (high dose) hematopoietic growth factors.
Time Frame: From engraftment to 60 days post transplant
Measure: Median (Full Range); unit: days
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 49
days | 18 [18 to 38]

5. Secondary Outcome: 2-year Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the interval between day of transplant and day of death or disease progression.
Time Frame: First 25-35 days post transplant and then every 3 months for a maximum of 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 49
percentage of participants | 26 [15 to 39]

6. Secondary Outcome: 2-year Overall Survival
Description: Overall Survival (OS) is defined as the interval between day of transplant and day of death.
Time Frame: First 25-35 days post transplant and then every 3 months for a maximum of 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 49
percentage of participants | 33 [20 to 46]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of informed consent, first 25-35 days post transplant and then every 3 months up to 2 years.
Arm/Group | Busulfan + Fludarabine + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 39/56
Other Adverse Events (participants affected / at risk) | 54/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan + Fludarabine + Cyclophosphamide (N=56)
Death (General disorders) | 39 (39)
BK virus associated hemorrhagic cystitis (Infections and infestations) | 2 (2)
Cardio-renal syndrome (Cardiac disorders) | 1 (1)
Chronic GI GvHD (Gastrointestinal disorders) | 1 (1)
Chronic ocular GvHD (Eye disorders) | 1 (1)
Delayed engraftment due to Cytoxan (Immune system disorders) | 1 (1)
Elevated bilirubin due to Sepsis (Metabolism and nutrition disorders) | 1 (1)
Delayed Engraftment (Immune system disorders) | 1 (1)
Elevated alanine aminotransferase due to drug related (Metabolism and nutrition disorders) | 1 (1)
Elevated bilirubin due to drug related (Metabolism and nutrition disorders) | 1 (1)
GI GvHD (Gastrointestinal disorders) | 3 (3)
Graft Failure due to Relapsed MDS (Immune system disorders) | 1 (1)
Graft Failure due to micro-environment (Immune system disorders) | 1 (1)
Graft Failure due to Rejection (Immune system disorders) | 4 (4)
Hemorrhage due to low PLT (Vascular disorders) | 1 (1)
Infections Viral (Infections and infestations) | 2 (2)
Liver GvHD (Hepatobiliary disorders) | 3 (3)
Infections Bacterial (Infections and infestations) | 4 (5)
Infections Fungal (Infections and infestations) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neutropenic typhlitis (Gastrointestinal disorders) | 1 (1)
Presumed viral encephalitis (Infections and infestations) | 1 (1)
Primary Graft Failure (Immune system disorders) | 1 (1)
Presumed fungal pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Thrombocytopenia due to Valcyte (Blood and lymphatic system disorders) | 1 (1)
Skin GVHD (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan + Fludarabine + Cyclophosphamide (N=56)
Abdominal pain due to Doxycycline (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Allergic reaction due to Platelet transfusion (Immune system disorders) | 1 (1)
Allergic reaction due to Cell infusion (Immune system disorders) | 1 (1)
Altered mental status changes due to drug related (Nervous system disorders) | 6 (6)
Altered mental status changes due to ATG (Nervous system disorders) | 1 (1)
Altered mental status changes (Nervous system disorders) | 3 (3)
Atrial fibrilation due to dexamethasone (Cardiac disorders) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
BK virus associated hemorrhagic cystitis (Infections and infestations) | 24 (24)
Bone pain due to Neupogen (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Chronic ocular GvHD (Eye disorders) | 4 (4)
Chronic skin GvHD (Skin and subcutaneous tissue disorders) | 1 (1)
Chronic upper GI GvHD (Gastrointestinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 5 (5)
Demodex folliculitis (Infections and infestations) | 1 (1)
Dermatitis drug eruption vs GvHD (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 21 (22)
Dizziness due to Dilantin (Nervous system disorders) | 1 (1)
Dysphagia due to radiation treatment (Gastrointestinal disorders) | 1 (1)
Elevated alanine aminotransferase (Metabolism and nutrition disorders) | 6 (6)
Elevated alanine aminotransferase due to drug related (Metabolism and nutrition disorders) | 7 (7)
Elevated alkaline phosphatase (Metabolism and nutrition disorders) | 4 (4)
Elevated alkaline phosphatase due to drug related (Metabolism and nutrition disorders) | 4 (4)
Elevated bilirubin (Metabolism and nutrition disorders) | 9 (9)
Elevated bilirubin due to RBC transfusions (Metabolism and nutrition disorders) | 1 (1)
Elevated bilirubin due to drug related (Metabolism and nutrition disorders) | 4 (4)
Elevated lactate dehydrogenase due to Vancomycin (Metabolism and nutrition disorders) | 1 (1)
Engraftment syndrome (Immune system disorders) | 1 (1)
Fevers (General disorders) | 10 (10)
Fevers due to ATG (General disorders) | 19 (19)
Fevers due to Engraftment Syndrome (General disorders) | 1 (1)
Fevers due to Transfusion (General disorders) | 1 (2)
Fluid overload (Blood and lymphatic system disorders) | 17 (17)
Gastritis (Gastrointestinal disorders) | 1 (1)
Folliculitis (Infections and infestations) | 3 (3)
GI GvHD (Gastrointestinal disorders) | 9 (9)
GI bleed of undetermnined cause (Gastrointestinal disorders) | 1 (1)
Headaches (Nervous system disorders) | 3 (3)
Hemochromatosis (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage of undetermined etiology (Vascular disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Hypertension due to Tacrolimus (Cardiac disorders) | 1 (1)
Hypotension due to Norvasc (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infections Bacterial (Infections and infestations) | 36 (65)
Infections Fungal (Infections and infestations) | 5 (6)
Infections Viral (Infections and infestations) | 33 (51)
Line related deep vein thrombosis (Vascular disorders) | 4 (4)
Liver GvHD (Hepatobiliary disorders) | 6 (9)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 2 (2)
Myopathy due to Tramadol (Musculoskeletal and connective tissue disorders) | 1 (1)
Magnesium induced diarrhea (Metabolism and nutrition disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 48 (48)
Nausea (Gastrointestinal disorders) | 48 (49)
Nausea due to drug related (Gastrointestinal disorders) | 2 (2)
Nausea due to CMV infection (Gastrointestinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Neutropenic fevers (Infections and infestations) | 30 (30)
Oral GvHD (Gastrointestinal disorders) | 2 (2)
Ocular GvHD (Eye disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Propionibaterium acnes conjunctivitis (Eye disorders) | 1 (1)
Pruritus due to Bactrim (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Rash due to ATG (Skin and subcutaneous tissue disorders) | 3 (3)
Rash due to drug related (Skin and subcutaneous tissue disorders) | 5 (6)
Red cell dysplasia due to ABO incompatibility (Blood and lymphatic system disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Renal insufficiency due to Nephrotoxins (Renal and urinary disorders) | 3 (3)
Renal insufficiency due to Pyelonephritis (Renal and urinary disorders) | 1 (1)
Renal insufficiency due to Overt diuresis (Renal and urinary disorders) | 1 (1)
Renal insufficiency due to drug related (Renal and urinary disorders) | 9 (9)
Renal insufficiency due to Obstructive neuropathy (Renal and urinary disorders) | 1 (1)
Renal insufficiency due to Obstructive uropathy (Renal and urinary disorders) | 1 (1)
Renal insufficiency due to Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1)
Shortness of breath due to platelet transfusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Severe vulvar discomfort (Reproductive system and breast disorders) | 1 (1)
Skin GVHD (Skin and subcutaneous tissue disorders) | 25 (27)
Steroid-Induced Myopathy (Musculoskeletal and connective tissue disorders) | 3 (3)
Small bowel obstruction from pneumatosis coli (Gastrointestinal disorders) | 1 (1)
Steroid induced hyperglycemia (Metabolism and nutrition disorders) | 16 (16)
Suspected cGvHD (Immune system disorders) | 1 (1)
Suspected metabolic encephalopathy (Metabolism and nutrition disorders) | 1 (1)
Suspected migraine (Nervous system disorders) | 1 (1)
Suspected Ganciclovir induced diarrhea (Gastrointestinal disorders) | 1 (1)
Suspected engraftment syndrome (Immune system disorders) | 1 (1)
Ulcer (General disorders) | 1 (1)
Upper GI GvHD (Gastrointestinal disorders) | 9 (9)
Thrombocytopenia due to drug related (Blood and lymphatic system disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes